CLINICAL TRIAL: NCT02987140
Title: Understand Freezing of Gait in Parkinson's Disease: Behavioral Physiology and Clinical Application
Brief Title: Understand FoG in PD: Behavioral Physiology and Clinical Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 201606057RINA
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Parkinson's disease; freezing of gait; context-dependency; transcranial magnetic stimulation; visual cues
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PD+FoG (Experimental): PD patients with FoG
  Interventions: Behavioral: Clinical evaluations
- PD-FoG (Active Comparator): PD patients without FoG
  Interventions: Behavioral: Clinical evaluations
- Control (Active Comparator): age-matched non-disabled adults
  Interventions: Behavioral: Clinical evaluations

INTERVENTIONS:
Behavioral: Clinical evaluations — Participants will receive clinical evaluations, and practice the finger sequence task used to assess context-dependency along with EEG assessment. On the second day, the participants will receive the TMS assessment.

SUMMARY:
The overall goals of this proposed study are to investigate the behavioral and neurophysiological mechanisms of patients with Parkinson's disease (PD) experiencing freezing of gait (FoG). More specifically, we aim to determine the behavioral changes in context-dependency and changes in corticomotor excitability associated with FoG.

DETAILED DESCRIPTION:
Background: Freezing of gait (FoG) is a debilitating symptom for patients with Parkinson's disease (PD). FoG not only impairs walking but also significantly increase fall risks and decrease quality of life for patients with PD. Despite the critical consequences, the mechanisms associated with this phenomenon are not well understood.

Clinically, FoG often occurs when individuals with PD are approaching a narrow pathway or crossing a busy street. This observation leads to the hypothesis that FoG is associated with context-dependent motor performance, a phenomenon that an individual demonstrate poorer performance if the learned motor task is carried out in an unfamiliar context. Whether the occurrence of freezing episodes is a result of context-dependency has not been systematically investigated. Moreover, the changes in corticomotor excitability associated with FoG have not been well-established.

Objectives: The objectives of this proposal are to understand the behavioral and neurophysiological mechanisms of FoG. The specific aim is to examine the behavioral changes in context-dependency and changes in corticomotor excitability associated with FoG.

Methods: a total of 70 participants, including PD patients with FoG, PD patients without FoG, and age-matched non-disabled adults, will be recruited. The participants will undergo behavioral and neurophysiological examinations. Behavioral evaluations will include context-dependent motor performance, FoG, disease severity, and walking and balance functions. Transcranial magnetic stimulation and electroencephalogram will be used to measure corticomotor excitability of the participants. Analysis of variance (ANOVA) and regression analysis will be performed to compare and determine the relationship between FoG, behavioral outcomes, and corticomotor excitability. Statistical significance level is set at p < 0.05.

ELIGIBILITY:
Inclusion criteria:

* Individuals with Parkinson's disease
* Healthy control subjects

Exclusion criteria:

* unable to follow the instructions
* have other neurological diseases other than PD
* have pacemaker implanted in their body
* have a history of seizure
* have a family history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
New Freezing of Gait Questionnaire (NFOG-Q) | 30 mins
  The New Freezing of Gait Questionnaire (NFOG-Q) will be used to evaluate the freezing frequency and severity of the patients with PD. It composes of 3 parts; in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. PartⅡassesses the severity of FoG according to the frequency and duration of the freezing episodes, while PartⅢevaluates the impact of freezing on daily activities, such as walking. The reliability and internal consistency of the NFOG-Q have been well-established for patients with PD (Nieuwboer et al., 2009).
Context-dependent behavior | 40 mins
  A modified finger sequence task is specifically designed to evaluate context-dependent behavior for patients with PD. The participants will be instructed to put their index and middle fingers of both hands on a designated location of an enlarged key-board.
  The participants will first practice the three sequences for a total of 324 practice trials on the first day. Ten minutes and 24 hours after practice, to control for the medication status, the participants will be tested under the SAME and SWITCH conditions.With these 2 testing conditions, we will be able to calculate a variable called Switch Cost, which is the performance difference between the SWTICH and the SAME conditions normalized by the SAME condition [100% * (SWITCH - SAME)/SAME]. The Switch Cost will be used as an indicator of context-dependency.

SECONDARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale (UPDRS) | 30 mins
  The UPDRS contains 4 sections, and PartIIIwill be used in this study to evaluate the motor disturbances of patients with PD. Excellent internal consistency and validity has been established for UPDRS (Goetz et al., 2008).
Montreal Cognitive Assessment (MoCA) | 10 mins
  The MoCA evaluates several cognitive domains, including visuospatial processing, naming, short-term memory, digit forward and backward span, verbal fluency, abstract concept, counting, and orientation. The MoCA has been found to be a valid and reliable tool to screen for cognitive dysfunctions in patients with PD (Gill, Freshman, Blender, & Ravina, 2008).
The Stroop Color-Word test | 5 mins
  The Stroop Color-Word test involves congruent and incongruent conditions.The goal of the participants is to read out the ink color of the word, but not the color word name itself, as accurately and as soon as possible (Dubois et al., 2007; Ridley, Johnson, & Braisted, 1978).
10-Meter Walk Test (10MWT) | 5 mins
  10MWT assesses the walking ability of the participants. The participants will be instructed to walk in their comfortable walking speed and their fastest walking speed for 10 meters. Gait speed, stride length, and cadence will be calculated.
The Timed Up and Go (TUG) test | 5 mins
  The TUG evaluates the balance ability of the participants. The participants will be seated on a comfortable chair with hip and knee flexed at 90 Upon a 'Go' signal, the participants will stand up from the chair, walk 3 meters, turn around, and sit back down to the chair. The time to complete the procedure will be measured.
The Parkinson's Disease Questionnaire(PDQ-39) | 10 mins
  The PDQ-39 specifically assess quality of life in patients with PD. PDQ-39 contains 39 questions embedded in 8 different domains. PDQ-39 has now become the most widely accepted and reliable measure to determine the overall health status for patients with PD (Jenkinson, Peto, Fitzpatrick, Greenhall, & Hyman, 1995).
Transcranial magnetic stimulation | 45 mins
  To compare the neurophysiological characteristics of PD patients with FoG, PD patients without FoG, and non-disabled adults, a TMS device (The Magstim Company Ltd, Whitland, UK) will be used. TMS outcomes will include resting motor threshold (RMT), motor evoked potentials (MEPs), cortical silent period (CSP), short-interval intracortical inhibition (SICI), long-interval intracortical inhibition (LICI), and intracortical facilitation (ICF).
Electroencephalogram (EEG) | 40 mins
  While performing the modified finger sequence task, the electroencephalogram (EEG) will be used to monitor and record brain activity. Comparisons will be made between the first block of practice, last block of practice, and the two testing conditions.
The short FoG and festination assessment score | 20 mins
  The short FoG and festination assessment score, developed by Ziegler and colleagues (2010), will be used to clinically assess freezing and festination episodes over a short time course. The participants will initially sit on a chair for 30 seconds, then they will be instructed to stand up and walk to a floor mark with 40 radius and make 360 turn clockwise and counter-clockwise. Then, the participants will walk through a door, turn around and walk back to the chair. The participants will be required to walk in a fast but safe speed. This evaluation approach has been demonstrated to be feasible and reliable for assessing the severity of freezing and festination.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Yun Lee, PHD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan